CLINICAL TRIAL: NCT01675206
Title: Randomized Prospective Open Interventional Multi-centre Study on Finding the Optimal Dose of Vitamin K2 Supplements for Hemodialysis Patients
Brief Title: Dose Defining Study for the Administration of Vitamin K2 Supplements in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rogier Caluwe (Other)
Responsible Party: Sponsor-Investigator, Rogier Caluwe, MD, Onze Lieve Vrouw Hospital
Organization: Onze Lieve Vrouw Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/066
Record Dates: First submitted 2012-08-22; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Vascular Calcification
Keywords: Vascular calcification; Hemodialysis; Matrix Gla Protein; Vitamin K2
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 360 µg Vit K2 (Active Comparator): Administration of 360 µg of Vitamin K2 thrice weekly
  Interventions: Dietary Supplement: Vitamin K2 supplementation
- 720 µg Vit K2 (Active Comparator): Administration of 720 µg of Vitamin K2 thrice weekly
  Interventions: Dietary Supplement: Vitamin K2 supplementation
- 1080 µg Vit K2 (Active Comparator): Administration of 1080 µg of Vitamin K2 thrice weekly
  Interventions: Dietary Supplement: Vitamin K2 supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin K2 supplementation

SUMMARY:
This study aims at finding the optimal dose of Vitamin K2 supplementation in hemodialysis patients.

DETAILED DESCRIPTION:
During the past few years evidence is emerging for a role of Matrix Gla Protein (MGP) as one of the most powerful inhibitors of vascular calcification (Shurgers LJ et al. Thromb Haemost 2008; 100: 593-603). MGP is a Vitamin K dependent protein. This means that he presence of Vitamin K2 is required to promote the gamma-carboxylation process turning MGP in its carboxylated and active form. Recent data show that dp-uc MGP correlates well with Vitamin K status (Cranenburg CM et al. Thrombosis and Haemostasis 2010; 104/4: 811-822).

It is widely recognized that patients with renal insufficiency treated with hemodialysis are prone to accelerated vascular calcification resulting in excess cardiovascular morbidity and mortality (Goodman WG et al. N Engl J Med 2000; 342: 1478-1483).

Consequently, the administration of Vitamin K2 supplements may protect hemodialysis patients against accelerated vascular calcification by enhancing the gamma-carboxylation process of MGP. However, the optimal dose of Vitamin K2 required to achieve these results remains to be defined

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 year
* signed informed consent
* end stage renal disease treated with chronic hemodialysis at least three times a week

Exclusion Criteria:

* coumarin treatment
* known intestinal malabsorption
* inability to take oral medication
* medical conditions with a considerable probability for death within 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
percentage of reduction in dp-ucMGP after 8 weeks of Vitamin K2 supplementation | 8 weeks
  this study aims at verifying whether higher doses of Vitamin K2 supplementation result in an increased reduction in dp-ucMGP

SECONDARY OUTCOMES:
Assessment of adverse reactions associated with Vitamin K2 intake | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rogier Caluwé, MD, Principal Investigator — OLV Hospital Aalst Belgium; Bruno Van Vlem, MD, PhD, Study Chair — OLV Hospital Aalst Belgium; An Devriese, MD, PhD, Study Chair — AZ St.-Jan Brugge Belgium; Stefaan Vandecasteele, MD, PhD, Study Chair — AZ St.-Jan Brugge Belgium